CLINICAL TRIAL: NCT04844411
Title: A Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-67835989 in Healthy Participants
Brief Title: A Study of JNJ-67835989 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108974; 2021-000337-14 (EudraCT Number); 67835989EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: JNJ-67835989 (Oral Suspension) (Experimental): Participants will receive a single oral suspension dose of JNJ-67835989 on Day 1 in Part 1 and Part 2.
  Interventions: Drug: JNJ-67835989
- Arm B: Placebo (Placebo Comparator): Participants will receive a single oral solution placebo on Day 1 in Part 1 only (except food effect cohorts).
  Interventions: Drug: Placebo
- Arm C: JNJ-67835989 (Oral Solid Dose) (Experimental): Participants will receive a single oral solid dose (tablet) of JNJ-67835989 on Day 1 in Part 3.
  Interventions: Drug: JNJ-67835989

INTERVENTIONS:
Drug: JNJ-67835989 — JNJ-67835989 will be administered orally.
  Arms: Arm A: JNJ-67835989 (Oral Suspension); Arm C: JNJ-67835989 (Oral Solid Dose)
Drug: Placebo — Matching placebo will be administered orally.
  Arms: Arm B: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of JNJ-67835989 versus placebo after single (or divided) oral dose administration (ascending dose levels) in healthy participants, pharmacokinetics (PK) of JNJ-67835989 in plasma and urine after single (or divided) oral dose administration in healthy participants, effects of JNJ-67835989 following single (or divided) oral dose administration in healthy participants on cardiovascular parameters, effects of JNJ-67835989 following single (or divided) oral dose administration on dissociative symptoms in healthy participants, and sedative effects of JNJ-67835989 following single (or divided) oral dose administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical and neurological examination, medical history, vital signs and 12-lead electrocardiogram (ECG) performed at screening. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable. The presence of complete Left Bundle Branch Block (LBBB), atrioventricular (AV) block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator (ICD) will lead to exclusion. Heart rate must be less than or equal to (<=) 90 beats per minute (bpm)
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, including liver enzymes, blood coagulation, hematology, thyroid function or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body mass index (BMI) within the range 18.0 and 29.9 kilograms per meter square (kg/m^2) (inclusive)
* A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person. Male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak
* Must sign an informed consent form (ICF) indicating that he understands the purpose of, and procedures required for, the study and is willing to participate in the study. Participation in the pharmacogenomic part of the study is mandatory
* Willing and able to adhere to the lifestyle restrictions specified in this protocol
* Part 2 only: Participants should be moderate to heavy cigarette smokers (at least 10 cigarettes per day; no e-cigarettes or cigars) for at least the 3 months prior to screening. Smoking will be allowed at specific times each day during the study as defined by site staff. Participants should continue their smoking behavior during the complete study period until at least after the follow-up visit

Exclusion Criteria:

* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hypertension, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, parkinson's disease, psychiatric disorders, infection, or any other illness that the investigator considers should exclude the participant
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin, or malignancy that in the opinion of the investigator, with written concurrence with the safety responsible physician, is considered cured with minimal risk of recurrence)
* Systolic blood pressure greater than (>)140 millimeters of mercury (mmHg), diastolic blood pressure >90 mmHg or respiratory rate > 18 at screening
* Has had coronavirus disease (COVID) as confirmed by a positive severe acute respiratory syndrome coronavirus-2 (SARS-COV-2) test (polymerase chain reaction [PCR] or rapid antigen test, not an antibody test) within the past 3 months and/or has required hospitalization for treatment of COVID at any timepoint and/or has reported sequelae from COVID at screening
* Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 30 days (or 5 half-lives whichever is longest) before the planned first dose of study intervention or is currently enrolled in an investigational study
* For Parts 1 and 3 only: Smokes cigarettes (or equivalent) and/or has used nicotine-based products within 3 months prior to screening
* For Parts 1 and 3 only: Positive urine cotinine dipstick test at screening or admission

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Abnormalities in Vital Signs | Up to 6 weeks
  Number of participants with abnormalities in vital signs (heart rate [HR], systolic blood pressure [SBP], diastolic blood pressure [DPB]), respiratory rate, pulse oximetry and temperature will be reported.
Number of Participants with Clinically Significant Clinical Laboratory Abnormalities | Up to 6 weeks
  Number of participants with clinically significant clinical laboratory abnormalities (chemistry, hematology, urinalysis) will be reported.
Number of Participants with Adverse Events (AEs) | Up to 6 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Abnormalities in Electrocardiogram (ECG) | Up to 6 weeks
  Number of participants with abnormalities in ECG will be reported.
Plasma Concentrations of JNJ-67835989 and Possible Metabolites | Predose, up to 48 hours post dose (up to Day 3)
  Plasma samples will be analyzed to determine concentrations of JNJ-67835989 and possible metabolites using a validated, specific, and sensitive liquid chromatography-tandem mass spectrometry (LC MS/MS) method.
Urine Concentrations of JNJ-67835989 and Possible Metabolites | Predose, up to 72 hours post dose (up to Day 4)
  Urine samples will be analyzed to determine JNJ-67835989 and possible metabolites concentrations using a qualified research LC-MS/MS method.
Number of Participants with Clinician-Administered Dissociative States Scale (CADSS) Score | Up to Day 1
  CADSS is an instrument for the measurement of present-state dissociative symptoms and will be administered to assess treatment-emergent dissociative symptoms. CADSS consists of 23 subjective items, divided into 3 components: depersonalization (items 3 to 7, 20, and 23), derealization (items 1, 2, 8 to 13, 16 to 19, and 21) and amnesia (items 14, 15, and 22). The participants responses are coded on a 5-point scale (from 0 equals to [=] not at all to 4=extremely). The total score is sum of the 23 items and range from 0 to 92 - best is 0 and worst is 92.
Number of Participants with Modified Observer's Assessment of Alertness/Sedation Scale (MOAA/S) Scores | Up to Day 1
  The MOAA/S will be used to measure treatment-emergent sedation, with correlation to levels of sedation defined by the American Society of Anesthesiologists (ASA) continuum. The MOAA/S scores range from 0=no response to painful stimulus (corresponds to ASA continuum for general anesthesia) to 5=readily responds to name spoken in normal tone (awake; corresponds to ASA continuum for minimal sedation).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency